CLINICAL TRIAL: NCT03354468
Title: The Effects of a Fall Prevention Program on Falls, Patient Safety Culture and Patient-perceived Safety. Two Cross-sectional Studies in Two Orthopedic Departments
Brief Title: The Effects of a Fall Prevention Program on Falls, Patient Safety Culture and Patient-perceived Safety
Status: Completed | Type: Observational
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Norwegian University of Science and Technology (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/2469
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Hospitalized Patients; Accidental Falls
Keywords: Prevention and Control; Patient Safety; Aged; Risk Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- fall prevention program time 1: orthopedic department in Kristiansund hospital before implementation of a fall prevention program
  Interventions: Behavioral: fall prevention program
- no fall prevention program time 1: orthopedic department in Ålesund hospital without fall prevention program
- fall prevention program time 2: orthopedic department in Kristiansund hospital after implementation of a fall prevention program
  Interventions: Behavioral: fall prevention program
- no fall prevention program time 2: orthopedic department in Ålesund hospital without fall prevention program

INTERVENTIONS:
Behavioral: fall prevention program — fall prevention program in orthopedic department, consisting of 1) Seven examples of risk factors which might cause falls (diseases and medications, movement, cognitive behavior, vision, continence, nutrition, and the room and surroundings), 2) Methods to detect the risk factors, and 3) Measures to avoid falls or protect the patient in case of a fall.
  Groups: fall prevention program time 1; fall prevention program time 2

SUMMARY:
The incidence of fractures in Norway is among the highest in the world, and falls are the sixth major contributor to years lived with disability. In elderly, a large part of 900 deaths from unintentional injuries per 100000 inhabitants per year, are due to falls and fractures. Fractures, especially hip fractures among the elderly, often result in pain, ailments, and reduced quality of life. In Norway, 11 % of all reports from the specialized health services were incidents related to falls. Worldwide, falls are among the most commonly reported adverse events in hospitals with prevalence rates in the order of 10 per 1000 patient days or 5-15 % of the patients, and are associated with both minor and major injuries. The results of preventive measures are conflicting.

In January 2011, the Norwegian health minister launched a national patient safety campaign called "In Safe hands". The campaign had three aims: 1) Reduce patient related adverse events, 2) Build sustainable systems and structures for patient safety, and 3) Improve the patient safety culture. Hospitals and primary care units were invited to participate in 16 specific and measurable areas for improvement. One out of four orthopedic departments at Møre og Romsdal Hospital Trust, Norway participated actively in a fall prevention program.

This study compares the changes in fall rates, the employees' perceived patient safety culture and the patient experienced safety before and after implementation of the fall prevention program at the orthopedic department in one hospital in the Møre & Romsdal Hospital Trust, and at the same time points i another hospital in the same Trust but not having implemented the program.

DETAILED DESCRIPTION:
The interventions are multifaceted and include short and long-term activities to prevent falls. Fall screening, performed with the Norwegian version of the risk assessment tool for falls in elderly "STRATIFY (score 0 - 5), is the main tool. In patients with a score of 2 or more, a comprehensive individual plan for fall prevention has been worked out for each patient with risk of fall, documented in the medical records, and communicated to the staff responsible for the patient. The plan includes practical initiatives like adjusting the beds, proper illumination, instructions not to leave the bed unaided, and appropriate shoes. There are also long-term measures like the treatment of underlying diseases, changes in medication associated with risk of fall, physical training, and healthier dietary habits. During the intervention, the process is measured and reported to the national campaign. The national intervention was designed for use in hospitals, care facilities and patients living at home. Most of the proposed activities aim at preventing falls in a long time perspective.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the orthopedic department at Kristiansund Hospital or Ålesund Hospital
* admitted during one the two registration periods: from November 1, 2011 to October 31, 2012; or from November 1, 2013 to October 31, 2014
* a stay in the hospital of at least 24 hours' duration

Exclusion Criteria:

* n.a.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study included all patients above 64 years of age admitted to the orthopedic departments at Kristiansund Hospital and Ålesund Hospital during the two registration periods from November 1, 2011 to October 31, 2012; and from November 1, 2013 to October 31, 2014 and with a stay in the hospital of at least 24 hours' duration.
Sampling Method: Non-Probability Sample
Enrollment: 3143 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
proportion of fallers during the registration period | 1 year registration period

CONTACTS AND LOCATIONS:
Overall Officials: Espen Remme, Study Director — Helse Møre og Romsdal HF
Locations (2):
- Norway (2):
  - Dept of Orthopedics, Ålesund
  - Dept of Orthopedics, Kristiansund

REFERENCES:
- [Result] Royset B, Talseth-Palmer BA, Lydersen S, Farup PG. Effects of a fall prevention program in elderly: a pragmatic observational study in two orthopedic departments. Clin Interv Aging. 2019 Jan 15;14:145-154. doi: 10.2147/CIA.S191832. eCollection 2019. PMID 30697039